CLINICAL TRIAL: NCT02512666
Title: Non Invasive Optical Imaging of Capillaries Through the Nailfold for White Blood Cell Enumeration in Patients With Hematologic Malignancies
Brief Title: Non Invasive Optical Imaging of WBC Count
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yi-Bin A. Chen, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 15-070
Record Dates: First submitted 2015-07-28; First posted 2015-07-31 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Hematologic Malignancy
Keywords: Hematologic malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non-Invasive Imaging (Experimental): Commercial portable optical microscope (AM4113-N5UT Dino-Lite ) which will be employed during the study for a pre determined time of non-invasive imaging of the nailfold capillaries in ASCT patients.
  For Autologous Stem Cell Transplant (ASCT) participants, the imaging will be performed once prior to ASCT upon admission to the hospital, and then daily after ASCT (starting on day +7) until count recovery
  Interventions: Device: AM4113-N5UT Dino-Lite

INTERVENTIONS:
Device: AM4113-N5UT Dino-Lite

SUMMARY:
This research study is looking at a small device that measures white blood cell (WBC) counts by being placed against the finger nail for participants who are undergoing stem cell transplantation at Massachusetts General Hospital or have a hematologic malignancy and are being seen as an outpatient.

DETAILED DESCRIPTION:
The objective of this study is to obtain data that would support the use of a method to obtain WBC counts from images of small blood vessels called capillaries. These would be obtained by pressing a small device on the surface of participants' finger nails to look through the nail. These images will be obtained using a portable microscope called the Dino-Lite Digital Microscope.

Having a non-invasive way to quickly measure WBC counts could be useful for a variety of healthcare applications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lymphoid malignancies or plasma cell dyscrasias who are admitted to the Massachusetts General Hospital to undergo autologous stem cell transplantation or are seen in the outpatient clinic
* Age ≥ 18 years
* Ability to understand and the willingness to sign a written informed consent document.
* Patients must have WBC ≥ 3000 / µl and ANC ≥ 1500 / µl at admission or their last clinical visit to be enrolled.

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition of baby oil.
* Myelodysplasia
* Skin phototype < 4 in the Fitzpatrick scale.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-09; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Video of nail-fold imaging captured by capillaroscope | 4 weeks
  Image acquisition from device to then analyze and compare with complete blood counts measured in a standard fashion

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Bin A Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data